CLINICAL TRIAL: NCT05182658
Title: The Use of Empagliflozin in Patients With Hypertrophic Cardiomyopathy
Brief Title: Empagliflozin in Hypertrophic Cardiomyopathy
Acronym: EMPA-REPAIR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Medical University of Bialystok (Other); University of Eastern Finland (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/ABM/01/00001
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-03

CONDITIONS: Hypertrophic Cardiomyopathy; Heart Failure
Keywords: Hypertrophic cardiomyopathy; Heart Failue; Empagliflozin; Sodium-glucose transport protein 2 inhibitor; SGLT2 inhibitor
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin group (Active Comparator): Patients in the empagliflozin group will receive 10 mg of empagliflozin once daily for 12 months
  Interventions: Drug: Empagliflozin 10 MG
- Control group (Placebo Comparator): Patients in the control group will receive placebo once daily for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — The proposed intervention will be administration of empagliflozin at a standard dose of 10 mg daily for a period of 12 months. Patients with diagnosed diabetes will be excluded from the study. Patients (n = 250) will be randomized in a double-blind fashion to empagliflozin or placebo group.
  Other Names: Jardiance
  Arms: Empagliflozin group
Drug: Placebo — The proposed intervention will be administration of placebo for a period of 12 months. Patients (n = 250) will be randomized in a double-blind fashion to empagliflozin or placebo group.
  Arms: Control group

SUMMARY:
The proposed intervention will be administration of empagliflozin at a standard dose of 10 mg daily for a period of 12 months. Patients with diagnosed diabetes will be excluded from the study. Patients (n = 250) will be randomized in a double-blind fashion to empagliflozin or placebo group. The primary endpoint of the study will be the change in peak oxygen uptake (VO2 max) measured in a cardiopulmonary exercise test. VO2max is an objective indicator of physical performance and will be evaluated before and after empagliflozin or placebo treatment.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is the most common genetic disease of the myocardium. Conventionally, the incidence of this disease was estimated at 1: 500 people, but it is probably higher and amounts to about 1: 200 cases. In Poland, this gives 76,000 to 190,000 people. HCM is asymptomatic in some people. In others, it is associated with progressive left ventricular diastolic dysfunction due to myocardial hypertrophy and fibrosis, eventually leading to systolic dysfunction and progressive heart failure. Both heart failure with preserved left ventricular ejection fraction (LVEF) and reduced LVEF are inevitably associated with impaired physical function, often affecting young, professionally and socially active individuals. An additional significant problem in patients with HCM is arrhythmias leading to an increased risk of sudden death.

At present, for patients with HCM, there is no treatment available, which could inhibit the progression of the disease. The methods of treatment proposed so far, affecting the various pathogenic mechanisms of hypertrophic cardiomyopathy, have proved to be ineffective.

The aim of the project is therefore to seek a therapeutic solution for a disease for which standard medicine does not yet offer satisfactory solutions.

Empagliflozin is a reversible, potent and selective competitive inhibitor of sodium-glucose co-transporter-2 (SGLT2). It is the main transporter responsible for the reabsorption of glucose from the glomerular filtrate into the bloodstream. Its inhibition in people with type 2 diabetes leads to an increase in urinary glucose excretion and a decrease in its concentration in the blood. In the study in patients with type 2 diabetes and high cardiovascular risk, the use of empagliflozin was associated with a significant decrease in mortality and the number of hospitalizations due to heart failure. The mechanisms responsible for beneficial effects of empagliflozin are not fully understood. It is underlined that effects leading to a reduction of oxidative stress, improvement of diastolic function, inhibition of myocardial fibrosis and, what is important, improvement of myocardial energy status and reduction of cardiomyocyte calcium overload, increase of sarcoplasmic reticulum Ca2+ ATPase 2 (SERCA2) activity, which are important pathophysiological mechanisms of HCM, leading to progressive myocardial hypertrophy and the development of heart failure.

The proposed intervention will be administration of empagliflozin at a standard dose of 10 mg daily for a period of 12 months. Patients with diagnosed diabetes will be excluded from the study. Patients (n = 250) will be randomized in a double-blind fashion to empagliflozin or placebo group. The primary endpoint of the study will be the change in peak oxygen uptake (VO2 max) measured in a cardiopulmonary exercise test. VO2max is an objective indicator of physical performance and will be evaluated before and after empagliflozin or placebo treatment. Secondary endpoints will be a change in the maximum left ventricular wall thickness, left ventricular mass, parameters of diastolic dysfunction, severity of myocardial fibrosis and improvement of its energy status.

An important aspect of the study will be the genetic analysis of the study group. Data in both human and experimental studies indicate that the benefits of treatment may be dependent on the patient's genotype. The pathomechanisms of heart failure development differ depending on the mutation found and the prognosis of patients is the worst in the case of HCM phenocopies as well as in patients with pathogenic variants in sarcomeric genes. It is therefore justified to examine the genetic profile of the population being studied. For this purpose, next generation sequencing (NGS) with whole exome sequencing (WES) is planned. This will detect both known and unknown variants in the genes responsible for developing HCM. In addition, the investigators hypothesized that the beneficial cardiac effects of empagliflozin may be dependent on genes involved in the pathophysiology of diabetes, and a separate research task with the participation of a foreign partner (University of Eastern Finland) was devoted to this issue.

The investigators believe that the social benefit of the project is greater than its costs, giving the prospect of treating a disease for which modern medicine turns out to be insufficient. Preventing the development of heart failure among patients with HCM, apart from the benefit for the patients themselves, will also translate into economic benefits for the health care and the social systems

ELIGIBILITY:
Inclusion Criteria:

* written, voluntary informed consent to participate in the study
* diagnosis of hypertrophic cardiomyopathy
* age ≥ 18 years

Exclusion Criteria:

* refusal to consent to participate in the study
* diagnosis of diabetes
* patients with hypertrophic obstructive cardiomyopathy requiring interventional treatment (maximal LVOT gradient ≥ 50 mmHg), and who are in III-IV NYHA functional class, despite of the treatment with maximal tolerated doses
* refusal to consent to participate in the study
* diagnosis of diabetes
* patients with hypertrophic obstructive cardiomyopathy requiring interventional treatment (maximal LVOT gradient ≥ 50 mmHg), and who are in III-IV NYHA functional class, despite of the treatment with maximal tolerated doses
* ICD or cardiac pacemaker (for a group of patients in whom cardiac magnetic resonance study will be performed; n=100)
* planned implantation of cardiac resynchronization therapy (CRT of CRT-D) in the following 12 months
* life expectancy below 12 months
* pregnancy (currently or planned in the following 12 months)
* breast feeding
* age below 18 years
* recurrent genito-urinary tract infections in the past or currently
* urosepsis in the history
* Impaired renal function, defined as eGFR < 30 mL/min/1.73 m2 (CKD-EPI)cr or requiring dialysis,
* other contraindications to the use of empagliflozin
* musculo-skeletal or neurologic diseases that make it unable to perform cardiopulmonary exercise testing
* heart transplant recipient or listed for heart transplant
* implanted left ventricular assist device
* Any severe (obstructive or regurgitant) valvular heart disease expected to lead to surgery during the trial in the Investigator's opinion
* Acute decompensated HF (exacerbation of chronic HF) requiring intravenous (i.v.) diuretics, i.v. inotropes or i.v. vasodilators, or left ventricular assist device within 1 week from discharge to screening, and during screening period until randomization
* Atrial fibrillation or atrial flutter with a resting heart rate > 110 bpm documented by ECG at screeining
* Systolic blood pressure (SBP) ≥ 180 mmHg at randomization
* Symptomatic hypotension and/or a SBP < 100 mmHg at screeining or randomization
* Chronic pulmonary disease requiring home oxygen, oral steroid therapy or hospitalisation for exacerbation within 12 months, or significant chronic pulmonary disease in the Investigator's opinion, or primary pulmonary arterial hypertension
* Indication of liver disease, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) at screening
* Haemoglobin < 9 g/dl at screening
* Major surgery (major according to the investigator's assessment) performed within 90 days prior to screening, or scheduled major elective surgery (e.g. hip replacement ) within 90 days after screening
* Gastrointestinal (GI) surgery or GI disorder that could interfere with absorption of trial medication in the investigator's opinion
* Any documented active or suspected malignancy or history of malignancy within 2 years prior to screening, except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of uterine cervix or low risk prostate cancer
* History of ketoacidosis
* Patients who must or wish to continue the intake of any drug considered likely to interfere with the safe conduct of the trial
* Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s), or receiving other investigational treatment(s)
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial subject or unlikely to complete the trial
* Any other clinical condition that would jeopardise patients safety while participating in this trial, or may prevent the subject from adhering to the trial protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Change in peak VO2 measured in the cardiopulmonary exercise testing | 12 months
  Change in peak VO2 measured in the cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Secondary outcome: Change in peak VO2 measured in the cardiopulmonary exercise testing in patients with reduced left ventricular ejection fraction (EF <50%) | 12 months
  Change in peak VO2 measured in the cardiopulmonary exercise testing in patients with reduced left ventricular ejection fraction (EF <50%)

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Śpiewak, MD, PhD, Principal Investigator — National Institute of Cardiology, Department of Radiology, Magnetic Resonance Unit; Mariusz Kłopotowski, MD, PhD, Principal Investigator — National Institute of Cardiology, Department of Cardiology and Interventional Angiology; Karol Kamiński, Professor, Principal Investigator — Medical University of Bialystok, Department of Population Medicine and Lifestyle Diseases Prevention
Locations (2):
- Poland (2):
  - Medical University of Bialystok, Bialystok
  - National Institute of Cardiology, Warsaw

IPD SHARING:
Plan to Share IPD: No